CLINICAL TRIAL: NCT00394524
Title: Trial Between a Computer-Guided Intravenous Infusion Protocol Versus a Standard Insulin Infusion Algorithm in Medical ICU
Brief Title: Trial Between a Computer-Guided Insulin Infusion Protocol Versus a Standard Insulin Infusion Algorithm in Medical ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Sanofi (Industry); Grady Health System (Other); Piedmont Healthcare (Other); University of Tennessee (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, MD, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00021877; IRB 830-2005 (Other: Emory University)
Record Dates: First submitted 2006-10-31; First posted 2006-11-01 (Estimated); Results first posted 2013-09-30 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Diabetes or With New Hyperglycemia
Keywords: ICU; hyperglycemia; glucommander
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Computer assisted IV insulin infusion (Experimental): Subjects in this group will receive continuous intravenous (IV) Insulin Infusion using glucommander computer guided system. All patients in the study will receive Glulisine(Apidra R ) a rapid acting insulin approved by Food and Drug Administration (FDA)
  Interventions: Device: Glucommander
- Standard insulin infusion algorithm (Active Comparator): Subjects in this group will receive Insulin using Standard insulin infusion algorithm. All patients in the study will receive Glulisine(Apidra R ) a rapid acting insulin approved by Food and Drug Administration (FDA)
  Interventions: Other: Standard insulin infusion algorithm

INTERVENTIONS:
Device: Glucommander — Glucommander is a Computer-guided Intravenous (IV) insulin infusion protocol used for glycemic control in inpatients. This algorithm directs the administration of IV insulin in response to Blood Glucose (BG) measurement at the patient's bedside. In this study, the Glucommander program was loaded into a PalmOne (Zire 31, Tungsten E2 by Palm Inc.) handheld personal digital assistant (PDA) device. During the infusion, the nurse entered BG levels into the system and the computer recommended the insulin infusion rate and a variable time to check the next glucose testing. An alarm prompted the scheduled glucose check. The insulin infusion followed the formula: Insulin/Hour = Multiplier × (BG- 60).
  Arms: Computer assisted IV insulin infusion
Other: Standard insulin infusion algorithm — Standard insulin infusion Algorithm is a standard paper form insulin infusion algorithm. The algorithm is divided into four columns based on empirically determined insulin sensitivity. The first column was for the most insulin-sensitive patients, and the fourth column was for the most insulin resistant patients. The majority of patients are started in the algorithm 1 column. Insulin resistant patients, such as those receiving glucocorticoids or receiving >80 units of insulin per day as outpatients, started in the algorithm 2 column. The insulin infusion rate was determined by the patient's BG level and was measured hourly until the patient was stable and within the target range. If BG targets were not achieved and the BG had not decreased by at least 60 mg/dL in the preceding hour, the patient was moved to the next column.
  Arms: Standard insulin infusion algorithm

SUMMARY:
The study is a multicenter, prospective, open-label randomized study to compare the safety and efficacy of continuous insulin infusion (CII) via a computer-guided(Glucommander) and a standard paper form protocol among the patients hospitalized in a medical intensive care unit (ICU).

.

DETAILED DESCRIPTION:
Increasing evidence from observational studies in hospitalized patients with and without diabetes indicates that hyperglycemia is a predictor of poor outcome. Blood glucose control with intensive insulin therapy in patients with acute critical illness reduces the risk of multiorgan failure and systemic infection, and decreases short- and long-term mortality.

The use of intravenous insulin infusion is the preferred route of insulin administration for the management of diabetic subjects with diabetic ketoacidosis and nonketotic hyperosmolar state, intraoperative and postoperative care, the postoperative period following heart surgery and organ transplantation, acute myocardial infarction, stroke, and critical care illness. Some of these settings may be characterized by, or associated with, severe or rapidly changing insulin requirements, generalized patient edema, impaired perfusion of subcutaneous sites, requirement for pressor support, and/or use of total parenteral nutrition. In these settings, the intravenous route for insulin administration has been considered superior than the subcutaneous injection of split-mixed regimen of intermediate and regular insulin with respect to rapidity of effect in controlling hyperglycemia, overall ability to achieve glycemic control, and most importantly, preventing hypoglycemic episodes. Recently, several insulin infusion protocols have been reported in the literature; these algorithms and formulas, however, may be confusing and difficult to follow and may increase the risk of dosing errors. To facilitate patients care, insulin algorithms could be placed on a computer and used at the patient bedside to direct the nursing staff administering the intravenous insulin. The Glucommander is one of such computer-derived insulin infusion protocol which has been used successfully in over 5,802 patients with diabetes between 1984 and 1998. The study hypothesizes that management of inpatient hyperglycemia with a computer-guided intravenous infusion protocol will facilitate smoother glycemic control with a lower rate of hypoglycemic events than treatment following a standard insulin infusion algorithm in critically ill patients in medical the ICU. The study also aims to determine differences in glycemic control between treatment with a computer-guided intravenous infusion protocol (Glucommander) and a standard insulin infusion algorithm in critically ill patients in the ICU.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between the ages of 18 and 70 years admitted to a medical ICU
2. A known history of diabetes mellitus or with new hyperglycemia untreated or treated by diet, insulin therapy or with any combination of antidiabetic agents (sulfonylureas, metformin, thiazolidinediones).

   * Blood glucose greater than 120 mg/dl on ≥ 2 occasions for known, treated diabetics or greater than 140 mg/dl on ≥ 2 occasions for those with new hyperglycemia.
3. Subjects must have an admission blood glucose < 400 mg/dL, without laboratory evidence of diabetic ketoacidosis (serum bicarbonate < 18 milliequivalents/L or positive serum or urinary ketones).

Exclusion Criteria:

1. Subjects with acute hyperglycemic crises such as diabetic ketoacidosis (DKA) and hyperosmolar hyperglycemic state [38].
2. Patients with known HIV, severely impaired renal function (serum creatinine ≥3.0 mg/dl).
3. Patients with mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
4. Female subjects who are pregnant or breast feeding at time of enrollment into the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2006-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo E Umpierrez, MD, Principal Investigator — Emory University SOM/Grady Health System; Bruce Bode, MD, Study Director — Piedmont Hospital; Abbas E Kitabchi, PhD,MD, Study Director — University of Tennessee Health Science Center, Memphis; Irl B Hirsch, MD, Study Director — University of Washington
Locations (4):
- United States (4):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Piedmont Hopsital, Atlanta, Georgia
  - University of Tennessee Health Science Center, Memphis, Memphis, Tennessee
  - University of Washington, Seattle, Seattle, Washington

REFERENCES:
- [Result] Newton CA, Smiley D, Bode BW, Kitabchi AE, Davidson PC, Jacobs S, Steed RD, Stentz F, Peng L, Mulligan P, Freire AX, Temponi A, Umpierrez GE. A comparison study of continuous insulin infusion protocols in the medical intensive care unit: computer-guided vs. standard column-based algorithms. J Hosp Med. 2010 Oct;5(8):432-7. doi: 10.1002/jhm.816. PMID 20945468

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4 hospital centers between April 2006 and August 2008.
Pre-assignment Details: Of 160 enrolled, 80 were randomized to each group. Among the 80 subjects in glucommander group, 1 died prior to starting infusion and 2 were excluded because of meeting exclusion criteria for the protocol. Among 80 subject in standard group 1 withdrew consent prior to starting infusion and 3 met exclusion criteria. 153 were analyzed
Groups:
- Glucommander: continuous insulin infusion per Glucommander, a computer-guided device; dosage or rate of insulin per algorithm
- Standard Insulin Infusion: standard continuous insulin infusion with columnar algorithm; dosage or rate of insulin per algorithm
Period: Overall Study
Arm/Group | Glucommander | Standard Insulin Infusion
Started | 80 | 80
Completed | 77 | 76
Not Completed | 3 | 4
Not completed — Protocol Violation | 2 | 3
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Glucommander: insulin infusion per Glucommander
- Standard Insulin Infusion: standard insulin infusion with columnar algorithm
- Total: Total of all reporting groups
Arm/Group | Glucommander | Standard Insulin Infusion | Total
Number analyzed (Participants) | 77 | 76 | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 62 | 52 | 114
  >=65 years | 15 | 24 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (11) | 58.5 (13.4) | 58.15 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 37 | 70
  Male | 44 | 39 | 83
Region of Enrollment [Number; unit: participants]
  United States | 77 | 76 | 153

OUTCOME MEASURES:

1. Primary Outcome: Mean Blood Glucose (BG) in mg/dl Among Glucommander Group Compared to Standard Insulin Infusion
Description: Daily mean blood glucose concentrations during insulin infusion with the Glucommander and a standard paper form insulin infusion algorithm are measured every day up until 10 days and a mean values of these levels are calculated. The Mean blood glucose concentrations are measured once the target blood glucose levels are achieved after admission
Time Frame: First 10 days of ICU stay
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Glucommander | Standard Insulin Infusion
Number analyzed (Participants) | 77 | 76
mg/dl | 103.3 (8.8) | 117.3 (16.5)

2. Secondary Outcome: Number of Patients With Severe Hypoglycemia Episodes Among the Glucommander Group Compared to Standard Algorithm
Description: Severe hypoglycemia is defined as the blood glucose (BG) levels lower than 40 mg/dL. The number of patients enrolled among both groups with the reports of having the BG levels lower than 40 mg/dL are recorded for duration of 10 days
Time Frame: First 10 days of ICU stay
Measure: Count of Participants; unit: Participants
Groups:
- Computer Assisted IV Insulin Infusion: Subjects in this group will receive continuous intravenous (IV) Insulin Infusion using glucommander computer guided system. All patients in the study will receive Glulisine(Apidra R ) a rapid acting insulin approved by Food and Drug Administration (FDA)
  Glucommander: Glucommander is a Computer-guided Intravenous (IV) insulin infusion protocol used for glycemic control in inpatients. This algorithm directs the administration of IV insulin in response to Blood Glucose (BG) measurement at the patient's bedside. In this study, the Glucommander program was loaded into a PalmOne handheld personal digital assistant (PDA) device. During the infusion, the nurse entered BG levels into the system and the computer recommended the insulin infusion rate and a variable time to check the next glucose testing. An alarm prompted the scheduled glucose check. The insulin infusion followed the formula: Insulin/Hour = Multiplier × (BG- 60).
- Standard Insulin Infusion Algorithm: Subjects in this group will receive Insulin using Standard insulin infusion algorithm. All patients in the study will receive Glulisine(Apidra R ) a rapid acting insulin approved by Food and Drug Administration (FDA)
  Standard insulin infusion Algorithm is a standard paper form insulin infusion algorithm. The algorithm is divided into four columns based on empirically determined insulin sensitivity. The first column was for the most insulin-sensitive patients, and the fourth column was for the most insulin resistant patients. The majority of patients are started in the algorithm 1 column. Insulin resistant patients, such as those receiving glucocorticoids or receiving >80 units of insulin per day as outpatients, started in the algorithm 2 column. The insulin infusion rate was determined by the patient's BG level and was measured hourly until the patient was stable and within the target range.
Arm/Group | Computer Assisted IV Insulin Infusion | Standard Insulin Infusion Algorithm
Number analyzed (Participants) | 77 | 76
Participants | 3 | 4

3. Secondary Outcome: Mean Length of Intensive Care Unit (ICU) in Days Stay Among Glucommander Group Compared to Standard Insulin Infusion Group
Description: Mean number of days, the patients stayed in the intensive care unit are measured among glucommander group and standard insulin infusion group.
Time Frame: During ICU hospitalization, up to 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Glucommander | Standard Insulin Infusion
Number analyzed (Participants) | 77 | 76
days | 8.5 (7.6) | 13.4 (13.8)

4. Secondary Outcome: Mean Hospital Length of Stay in Days Among the Glucommander Group Compared to Standard Insulin Infusion
Description: mean number of days the patients stayed in the hospital are measured among the Glucommander group and standard insulin infusion and compared
Time Frame: During the complete length of hospitalization, up to 60 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Glucommander | Standard Insulin Infusion
Number analyzed (Participants) | 77 | 76
days | 23.9 (26.3) | 17.5 (15)

ADVERSE EVENTS:
Time Frame: Adverse events for this study are collected for the duration of patients stay (patient's discharge or death) in the hospital among the Glucommander group and standard insulin infusion group which is up to 60 days
Description: The study is a comparison study between two insulin infusion algorithms among the hospitalized patients. For this study, since the intervention involves maintaining the glucose levels per the methods that are already approved the adverse events of interest are hypoglycemia and hyperglycemia.
Arm/Group | Glucommander | Standard Insulin Infusion
All-Cause Mortality (participants affected / at risk) | 17/77 | 20/76
Serious Adverse Events (participants affected / at risk) | 3/77 | 4/76
Other Adverse Events (participants affected / at risk) | 42/77 | 41/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Glucommander (N=77) | Standard Insulin Infusion (N=76)
Severe Hypoglycemia (Endocrine disorders) | 3 | 4 — Severe Hypoglycemia is defined as blood glucose levels <40 mg/dL
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Glucommander (N=77) | Standard Insulin Infusion (N=76)
Mild Hypoglycemia (Endocrine disorders) | 33 | 23 — Mild hypoglycemia is defined as blood glucose level <60 mg/dL
Hyperglycemia (Endocrine disorders) | 9 | 18 — Hyperglycemia is defined as blood glucose level of >200 mg/dL

LIMITATIONS AND CAVEATS:
Study was conducted in the medical ICU and excluded postsurgical patients and subjects expected to undergo a major surgical procedure, patients with severe renal insufficiency and with a history of hyperglycemic crises.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No